CLINICAL TRIAL: NCT01063569
Title: Glucocorticoid Treatment in Addison's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3.2007.2343; 2009-010917-61 (EudraCT Number)
Record Dates: First submitted 2010-01-26; First posted 2010-02-05 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Addison's Disease
Keywords: Addison's disease; Glucocorticoid treatment; Continuous subcutaneous hydrocortisone infusion; CSHI; Quality of Life; Sleep
MeSH Terms: conditions — Addison Disease | interventions — hydrocortisone hemisuccinate; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral hydrocortisone (Active Comparator)
  Interventions: Drug: Cortef (hydrocortisone)
- Continous subcutaneous hydrocortisone infusion (Experimental)
  Interventions: Drug: Solu-Cortef (hydrocortisone)

INTERVENTIONS:
Drug: Solu-Cortef (hydrocortisone) — Continuous Subcutaneous Hydrocortisone infusion via insulin pump. Doses adjusted to body surface area.
  Other Names: Solu-Cortef
  Arms: Continous subcutaneous hydrocortisone infusion
Drug: Cortef (hydrocortisone) — Oral treatment 3 times a day. Weight adjusted doses.
  Other Names: Cortef 5 mg
  Arms: Oral hydrocortisone

SUMMARY:
Addison's disease is a rare condition which in most cases is caused by autoimmune destruction of the adrenals, leading to deficiency of cortisol, aldosterone and adrenal androgens. Unrecognized the disease is life threatening, but with proper treatment patients can live near normal lives.

The conventional glucocorticoid replacement therapy renders the cortisol levels unphysiological, which may cause symptoms and long-term complications. Glucocorticoid replacement therapy is technically feasible by continuous subcutaneous hydrocortisone infusion (CSHI), and can mimic the normal diurnal cortisol rhythm. This study aims to further evaluate CSHI treatment in terms of metabolic effects, effects on health-related quality-of-life and sleep in an 8 months randomised open label clinical trial with crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with verified Addison's disease on stable treatment.

Exclusion Criteria:

* Insulin treated Diabetes Mellitus, cardiovascular disease,malignant disease, pregnancy.
* Treatment with glucocorticoids or drugs that interfere with cortisol metabolism (antiepileptics, rifampicin, St. John's wart).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Morning (08-09) plasma ACTH | Time 0, months 2, 3, 5, 7 and 8

SECONDARY OUTCOMES:
Health-Related Quality of Life; evaluated by SF-36 vitality scores and AddiQoL scores | At time 0 and months 2,3,5,7 and 8
Sleep; evaluated by Pittsburgh Sleep Quality Index (PSQI), and 7-days' Actigraph registration combined with self-reported sleep diary | PSQI: 0 and months 2,3,5,7 and 8; Actigraph/sleep diary: months 2 and 7
24h cortisol profiles in serum and saliva | months 2 and 7
S-glucose, 24 h profile | months 2 and 7
Insulin sensitivity assessed by euglycemic clamp | Months 2 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Løvås, MD,PhD, Principal Investigator — Haukeland University Hospital
Locations (3):
- Haukeland University Hospital, Bergen, Norway
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Uppsala University, Uppsala